CLINICAL TRIAL: NCT04988711
Title: Evaluation of the Reliability of a Non-invasive Tool for Measuring Hemoglobin in Severe Trauma Patients in the Emergency Room
Brief Title: Non-invasive Tool for Measuring Hemoglobin in Severe Trauma Patients in the ED
Acronym: HbOxymeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HbOxymeter
Record Dates: First submitted 2021-05-28; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: descriptive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hb Oxymeter (Experimental): Hb mesurment
  Interventions: Diagnostic Test: Hb Oxymeter

INTERVENTIONS:
Diagnostic Test: Hb Oxymeter — Measurement of Hb Oximeter

SUMMARY:
The development of miniaturized analytical technologies has facilitated the gradual decentralization of part of the laboratory examinations to the patient.

In addition, investigators are currently seeing the development of tools for non-invasive measurement of certain biological parameters. Thanks to their ease of use, results are obtained almost immediately and with good performance. These "rapid" tests or techniques should, in theory, reduce the time taken to take charge of patients, particularly in emergencies or in critical situations where the therapeutic decision should be as rapid and efficient as possible. These means, by their ease and speed of results, could be associated with the clinical examination of the practitioner to increase his diagnostic performance.

DETAILED DESCRIPTION:
It should be remembered that the journey of samples from the emergency room to the central laboratory, then the return of results is broken down into three phases: 1) the pre-analytical phase which includes medical prescription, sampling, request for analysis and delivery to 'at the central laboratory; 2) the analytical phase, specific to the laboratory, and which includes handling the sample and the analysis itself. This stage ends with the provision of the results (computer notification) and 3) the third stage (post analytical) represents the time between the provision of the results, their reading and their interpretation. All of these three phases constitute the recognized prescription-results-treatment time: Therapeutic Turn-around Time (TTAT). The main objective of these revolutionary techniques is to reduce this time or the duration of these three stages.

Several techniques, in particular delocalized biology, have been evaluated and validated in emergencies or even at home. In addition, non-invasive means remain underestimated in terms of relevance and reliability, mainly by lack of evaluation.

These measurement techniques relocated to the patient's bed allow rapid, non-invasive measurement without the need for intravenous access or the need to draw venous, arterial or capillary blood. These non-invasive devices can be portable, inexpensive, easy to use, and offer great benefits especially in emergency departments and pre-hospital settings. The accuracy of these methods is acceptable in the stable ICU patient. But that remains unassessed in an emergency.

Pulse co-oximetry or low perfusion oximetry is one of these technological advances being designed to allow the measurement of hemoglobin in a non-invasive manner. In addition, the automated spectrophotometric detection technique from a blood sample represents the Gold standard for the measurement of hemoglobin and has been recommended for several decades by the International Committee for Standardization in Hematology. This technique, performed in a hematology laboratory, allows precise, reliable and reproducible measurement. However, it requires a blood sample and above all imposes an incompressible delay. This dosage is one of the most prescribed samples in current practice in the emergency room. The possibility of determining the hemoglobin concentration in the patient's bed and non-invasively is a very attractive solution for the emergency physician.

The value of such a technique in trauma pathology seems indisputable. In fact, injuries represent a major problem for public health, representing more than 9% of deaths in the world each year. In particular, post-traumatic hemorrhage is the most common cause of preventable deaths, accounting for 50% of preventable deaths in the first 24 hours after major trauma. Early detection of hypovolaemia due to hemorrhage can be difficult, but essential for the patient's prognosis through an appropriate and adapted transfusion strategy. The hemoglobin dosage is essential for the emergency physician. Therefore, in the hospital setting, there is growing interest in rapid techniques for measuring hemoglobin.

Recently, a new device, Pronto-7, a point-controlled pulse CO-oximeter, has been developed. The Pronto-7 Spot Check Pulse CO-Oximeter has a spectrophotometric sensor (Rainbow DCI) that detects multiple wavelengths of light. The pulse CO-oximetry method discerns the distinctive light absorption characteristics of different hemoglobin species and applies proprietary algorithms to determine hemoglobin levels.

Few studies have investigated the effectiveness of this non-invasive hemoglobin measurement tool in trauma patients. No study in Tunisia has looked at the validation of this tool in terms of reliability, hence the interest of this study.

ELIGIBILITY:
Inclusion Criteria:

* Severe trauma patients
* Patients having benefited from a blood sample to measure hemoglobin.

Exclusion Criteria:

* Patients less than 3 years old.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | during the intervention
  The accuracy of Hb Oxymeter
the impact Hb Oxymeter | during the intervention
  the impact Hb Oxymeter

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (2):
- Tunisia (2):
  - HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul
  - Riadh Boukef, Sahloul, Sousse Governorate

IPD SHARING:
Plan to Share IPD: No
all data will be presented in the article publication